CLINICAL TRIAL: NCT00804570
Title: A Phase 2 Study of LY2196044 Compared With Placebo in the Treatment of Alcohol Dependence
Brief Title: A Study for the Treatment of Alcohol Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11359; H9T-MC-NABJ (Other: Eli Lilly and Company)
Record Dates: First submitted 2008-12-05; First posted 2008-12-09 (Estimated); Results first posted 2017-02-03 (Estimated); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Alcohol Dependence
MeSH Terms: conditions — Alcoholism | interventions — LY2196044

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- LY2196044 (Experimental)
  Interventions: Drug: LY2196044
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: LY2196044 — 250 milligram (mg) (titrate via 1 week at 50 mg and 1 week at 125 mg), once daily, orally, 16 weeks
  Arms: LY2196044
Drug: placebo — once daily, orally, 16 weeks
  Arms: Placebo

SUMMARY:
The Primary objective of this study is to test whether LY2196044 can reduce the number of heavy drinking days per month in people with alcohol dependence. Each subject will undergo a screening and assessment period (including medication washout) prior to randomization into a 16 week double blind treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Have Alcohol Dependence. Subjects must manifest at least the following 3 requirements for their diagnosis of Alcohol Dependence:

  1. Be tolerant, as defined by either of the following:

     1. A need for markedly increased amounts of alcohol to achieve intoxication or desired effect.
     2. Markedly diminished effect with continued use of the same amount of alcohol.
  2. Consume alcohol, often in larger amounts or over a longer period than was intended.
  3. Have a persistent desire or unsuccessful effort(s) to reduce or control alcohol use.
* Drink on average more than 14 drinks (women) or 21 drinks (men) per week with at least 2 heavy drinking days per week (≥4 drinks/day for women and ≥5 drinks/day for men) during the consecutive 30 day period prior to Screening and maintained through Randomization.
* Endorse abstinence or reduction in drinking.
* Female subjects of childbearing potential must have a negative urine pregnancy test and agree to use a reliable method of birth control during the study and for 2 months following the last dose of study drug.

Exclusion Criteria:

* Have experienced an acute alcohol withdrawal syndrome within the past 6 months or are currently at significant risk of suffering an acute alcohol withdrawal syndrome.
* Have a history of serious head injury, intracranial neoplasm or hemorrhage, prior seizure (other than remote history of childhood febrile seizure), or other condition that would place the subject at increased risk of seizure.
* Have ever taken anticonvulsants for seizure control.
* Are diagnosed with substance dependence or abuse (other than alcohol, cannabis, nicotine, or caffeine) within 6 months prior to Screening.
* Are receiving intensive behavioral or psychological therapy, delivered by a licensed or certified alcohol treatment specialist, for alcohol dependence.
* Meet criteria for a lifetime diagnosis of Schizophrenia, Schizoaffective Disorder, Bipolar I Disorder, or other psychoses.
* Have signs and symptoms of an active illness within the past 6 months of Screening for a diagnosis of Major Depressive Disorder (MDD) or Anxiety Disorder, or have a Cognitive Disorder diagnosed by clinical assessment. Subjects who were diagnosed with MDD in the more distant past, but have had a recent diagnosis of an active Major Depressive Episode, will not be eligible.
* Are actively suicidal, in the opinion of the investigator.
* Have taken any opiate or opioid analgesic (for example, codeine, hydrocodone) or an opiate receptor antagonist (for example, naltrexone) within 14 days prior to Screening.
* Are currently taking any medication excluded by the protocol.

  * Note: Subjects who discontinue/washout excluded medications prior to Randomization are not excluded from participation.
* Have evidence of significant active cardiac, respiratory, renal, gastrointestinal, or hematologic disease.
* Have acute or active hepatitis or hepatic inflammation.
* Have a history of cirrhosis or laboratory evidence of significant hepatocellular injury.
* Have plasma levels of sodium, potassium, calcium, magnesium, or phosphorous that fall outside of established reference ranges of the central laboratory for those analytes [that is, below lower limit of normal (LLN) or above upper limit of normal (ULN)] unless corrected prior to randomization.
* Have electrocardiogram (ECG) abnormalities obtained at Screening that are clinically significant with regard to the subject's participation in the study.
* Are women who are either pregnant or breast feeding.
* Have received treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry.
* Have previously completed or withdrawn from this study or any other study investigating LY2196044.
* Are unable, unreliable, and/or unwilling to provide informed consent, make themselves available for the duration of the study or abide by study procedures and restrictions.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Actual)
Dates: Start 2008-11; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (17):
- United States (17):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lafayette, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baltimore, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Belmont, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rochester, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Omaha, Nebraska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lebanon, New Hampshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New York, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chapel Hill, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charlotte, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cincinnati, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Portland, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Providence, Rhode Island
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charleston, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LY2196044 | Placebo
Started | 187 | 188
Completed | 115 | 94
Not Completed | 72 | 94
Not completed — Adverse Event | 14 | 7
Not completed — Lack of Efficacy | 0 | 1
Not completed — Lost to Follow-up | 18 | 21
Not completed — Entry criteria not met | 5 | 5
Not completed — Protocol Violation | 12 | 16
Not completed — Physician Decision | 1 | 2
Not completed — Sponsor decision | 1 | 4
Not completed — Withdrawal by Subject | 21 | 38

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LY2196044 | Placebo | Total
Number analyzed (Participants) | 187 | 188 | 375
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.92 (10.62) | 44.79 (10.08) | 44.85 (10.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 66 | 132
  Male | 121 | 122 | 243
Race/Ethnicity, Customized [Number; unit: participants]
  White | 152 | 134 | 286
  Black or African American | 26 | 43 | 69
  Asian | 1 | 1 | 2
  American Indian or Alaska Native | 0 | 3 | 3
  Multiple races | 7 | 7 | 14
  Unknown/Missing | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 187 | 188 | 375
Years of Alcohol Use [Mean (Standard Deviation); unit: years] | 30.64 (9.50) | 28.60 (10.44) | 29.53 (10.02)
Years of Heavy Drinking [Mean (Standard Deviation); unit: years] — Heavy drinking is defined as ≥4 drinks/day for women and ≥5 drinks/day for men.
  years | 25.06 (13.20) | 24.83 (11.00) | 24.94 (12.05)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Heavy Drinking Days at Week 16 Endpoint
Description: The Timeline Followback Method assesses the subject's daily drinking by means of a calendar that covers a specific time period and was used to assess the number of heavy drinking days. Heavy drinking is defined as ≥4 drinks/day for women and ≥5 drinks/day for men. Least Squares (LS) Mean value was controlled for treatment, pooled investigator, visit, gender, family history, treatment*visit, gender*family history, baseline, and baseline*visit. An unstructured covariance structure was used.
Time Frame: Week 16
Population: Participants with a baseline and post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: percentage of days
Arm/Group | LY2196044 | Placebo
Number analyzed (Participants) | 181 | 172
percentage of days | -43.02 (2.09) | -38.72 (2.12)
Statistical Analysis 1: Comparison: LY2196044 vs Placebo; Test type: Superiority or Other; p = 0.120, Mixed Models Analysis; Mean Difference (Final Values) = -4.30, 95% CI 2-sided [-9.72 to 1.13]

2. Secondary Outcome: Change From Baseline in Drinks Per Day at Week 16 Endpoint
Description: The Timeline Followback Method assesses the subject's daily drinking by means of a calendar that covers a specific time period and was used to assess the number of drinks consumed per day. Least Squares (LS) Mean value was controlled for treatment, pooled investigator, visit, gender, family history, treatment*visit, gender*family history, baseline, and baseline*visit. An unstructured covariance structure was used.
Time Frame: Baseline, Week 16
Population: Participants with a baseline and post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: number of drinks/day
Arm/Group | LY2196044 | Placebo
Number analyzed (Participants) | 185 | 179
number of drinks/day | -5.37 (0.22) | -4.66 (0.22)
Statistical Analysis 1: Comparison: LY2196044 vs Placebo; Test type: Superiority or Other; p = 0.013, Mixed Models Analysis; Mean Difference (Final Values) = -0.71, 95% CI 2-sided [-1.27 to -0.15]

3. Secondary Outcome: Change From Baseline in Percentage of Days Abstinent at Week 16 Endpoint
Description: The Timeline Followback Method assesses the subject's daily drinking by means of a calendar that covers a specific time period and was used to assess the percentage of days abstinent. Least Squares (LS) Mean value was controlled for treatment, pooled investigator, visit, gender, family history, treatment*visit, gender*family history, baseline, and baseline*visit. An unstructured covariance structure was used.
Time Frame: Baseline, Week 16
Population: Participants with a baseline and post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: percentage of days
Arm/Group | LY2196044 | Placebo
Number analyzed (Participants) | 181 | 172
percentage of days | 33.49 (2.05) | 28.12 (2.09)
Statistical Analysis 1: Comparison: LY2196044 vs Placebo; Test type: Superiority or Other; p = 0.051, Mixed Models Analysis; Mean Difference (Final Values) = 5.37, 95% CI 2-sided [-0.02 to 10.77]

4. Secondary Outcome: Change From Baseline in Drinks Per Drinking Day at Week 16 Endpoint
Description: The Timeline Followback Method assesses the subject's daily drinking by means of a calendar that covers a specific time period and was used to assess the number of drinks consumed on the days the participant drank. Least Squares (LS) Mean value was controlled for treatment, pooled investigator, visit, gender, family history, treatment*visit, gender*family history, baseline, and baseline*visit. An unstructured covariance structure was used.
Time Frame: Baseline, Week 16
Population: Participants with a baseline and post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: number of drinks/drinking day
Arm/Group | LY2196044 | Placebo
Number analyzed (Participants) | 182 | 178
number of drinks/drinking day | -3.77 (0.26) | -3.38 (0.26)
Statistical Analysis 1: Comparison: LY2196044 vs Placebo; Test type: Superiority or Other; p = 0.249, Mixed Models Analysis; Mean Difference (Final Values) = -0.40, 95% CI 2-sided [-1.07 to 0.28]

5. Secondary Outcome: Change From Baseline in Drinks Per Heavy Drinking Day at Week 16 Endpoint
Description: The Timeline Followback Method assesses the subject's daily drinking by means of a calendar that covers a specific time period and was used to assess the number of drinks consumed on heavy drinking days. Heavy drinking is defined as ≥4 drinks/day for women and ≥5 drinks/day for men. Least Squares (LS) Mean value was controlled for treatment, pooled investigator, visit, gender, family history, treatment*visit, gender*family history, baseline, and baseline*visit. An unstructured covariance structure was used.
Time Frame: Baseline, Week 16
Population: Participants with a baseline and post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: number of drinks/heavy drinking day
Arm/Group | LY2196044 | Placebo
Number analyzed (Participants) | 178 | 175
number of drinks/heavy drinking day | -2.61 (0.26) | -2.17 (0.26)
Statistical Analysis 1: Comparison: LY2196044 vs Placebo; Test type: Superiority or Other; p = 0.199, Mixed Models Analysis; Mean Difference (Final Values) = -0.44, 95% CI 2-sided [-1.12 to 0.23]

6. Secondary Outcome: Change From Baseline in Obsessive Compulsive Drinking Scale (OCDS) Total Score at Week 16 Endpoint
Description: Cravings will be assessed using the OCDS. The OCDS is a 14-item self-rating instrument. Total scores range from 0-40. Higher scores indicate more obsessive and craving. Least Squares (LS) Mean value was controlled for treatment, site, visit, gender, history, baseline, gender*history, treatment*visit, baseline*visit, gender*treatment, gender*treatment*visit. Subject was treated as a random effect. An unstructured covariance structure was used.
Time Frame: Baseline, Week 16
Population: Participants with a baseline and post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2196044 | Placebo
Number analyzed (Participants) | 174 | 162
units on a scale | -8.64 (0.51) | -7.96 (0.53)
Statistical Analysis 1: Comparison: LY2196044 vs Placebo; Test type: Superiority or Other; p = 0.318, Mixed Models Analysis; Mean Difference (Final Values) = -0.68, 95% CI 2-sided [-2.03 to 0.66]

7. Secondary Outcome: Change From Baseline in Drinker Inventory of Consequences (DrInC) - Recent Consequences (DrInC-2R) Total Score at Week 16 Endpoint
Description: DrInC is a self-administered, 50-item questionnaire designed to measure adverse consequences of alcohol abuse in 5 areas: Interpersonal, Physical, Social, Impulsive, and Intrapersonal. DrInC-2R provides a measurement since the last interview. Total scores range from 0-150, and higher scores indicate greater severity of symptoms. Least Squares (LS) Mean value was controlled for treatment, pooled investigator, visit, gender, family history, baseline, gender*family history, treatment*visit, baseline*visit. Subject was treated as a random effect. An unstructured covariance structure was used.
Time Frame: Baseline, Week 16
Population: Participants with a baseline and post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2196044 | Placebo
Number analyzed (Participants) | 148 | 136
units on a scale | -16.54 (1.09) | -13.53 (1.11)
Statistical Analysis 1: Comparison: LY2196044 vs Placebo; Test type: Superiority or Other; p = 0.034, Mixed Models Analysis; Mean Difference (Final Values) = -3.01, 95% CI 2-sided [-5.80 to -0.22]

8. Secondary Outcome: Ratio of Geometric Means Over Baseline in Gamma-Glutamyltransferase (GGT) Level at Week 16 Endpoint
Description: GGT and carbohydrate-deficient transferrin (%CDT) will be used as biochemical markers of alcohol consumption. A combination of GGT and %CDT improves the sensitivity of detecting excessive alcohol consumption as compared to either marker alone, or other traditional markers. Elevated levels indicate heavy alcoholism. Least Squares (LS) Mean value was controlled for treatment, pooled investigator, visit, gender, family history, baseline, gender*family history, treatment*visit, baseline*visit. An unstructured covariance structure was used.
Time Frame: Week 16
Population: Participants with a baseline and post-baseline value.
Measure: Geometric Mean (Standard Error); unit: ratio
Arm/Group | LY2196044 | Placebo
Number analyzed (Participants) | 176 | 161
ratio | 0.85 (0.02) | 0.94 (0.02)
Statistical Analysis 1: Comparison: LY2196044 vs Placebo; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis; GMR over Baseline relative to placebo = 0.90, 95% CI 2-sided [0.85 to 0.96]

9. Secondary Outcome: Ratio of Geometric Means Over Baseline in Percent Carbohydrate-Deficient Transferrin (%CDT) Level at Week 16 Endpoint
Description: Gamma-Glutamyltransferase (GGT) and %CDT will be used as biochemical markers of alcohol consumption. A combination of GGT and %CDT improves the sensitivity of detecting excessive alcohol consumption as compared to either marker alone, or other traditional markers. Elevated levels indicate heavy alcoholism. Least Squares (LS) Mean value was controlled for treatment, pooled investigator, visit, gender, family history, baseline, gender*family history, treatment*visit, baseline*visit. An unstructured covariance structure was used.
Time Frame: Week 16
Population: Participants with a baseline and post-baseline value.
Measure: Geometric Mean (Standard Error); unit: ratio
Arm/Group | LY2196044 | Placebo
Number analyzed (Participants) | 173 | 157
ratio | 0.90 (0.02) | 0.94 (0.02)
Statistical Analysis 1: Comparison: LY2196044 vs Placebo; Test type: Superiority or Other; p = 0.103, Mixed Models Analysis; GMR over Baseline relative to placebo = 0.96, 95% CI 2-sided [0.91 to 1.01]

10. Secondary Outcome: Ratio of Geometric Means Over Baseline in Aspartate Transaminase (AST) Level at Week 16 Endpoint
Description: AST is a potential biomarker for LY2196044 efficacy as decreases reflect decreased alcohol consumption. Least Squares (LS) Mean value was controlled for treatment, pooled investigator, visit, gender, family history, baseline, gender*family history, treatment*visit, baseline*visit. An unstructured covariance structure was used.
Time Frame: Week 16
Population: Participants with a baseline and post-baseline value.
Measure: Geometric Mean (Standard Error); unit: ratio
Arm/Group | LY2196044 | Placebo
Number analyzed (Participants) | 176 | 161
ratio | 0.88 (0.02) | 0.94 (0.02)
Statistical Analysis 1: Comparison: LY2196044 vs Placebo; Test type: Superiority or Other; p = 0.012, Mixed Models Analysis; GMR over Baseline relative to placebo = 0.94, 95% CI 2-sided [0.89 to 0.99]

11. Secondary Outcome: Change From Baseline in Beck Depression Inventory II (BDI-II) Total Score at Week 16 Endpoint
Description: The BDI-II contains 21 items that characterize how the subject was feeling in the past 2 weeks. There is a 4-point scale for each item ranging from 0 to 3 (0=no depression; 3=very depressed). Total scores range from 0-63. Higher scores indicate greater severity of depression. Least Squares (LS) Mean value was controlled for treatment, pooled investigator, gender, family history, baseline, gender*family history, treatment*visit, baseline*visit. An unstructured covariance structure was used.
Time Frame: Baseline, Week 16
Population: Participants with a baseline and post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2196044 | Placebo
Number analyzed (Participants) | 185 | 179
units on a scale | -3.10 (0.28) | -2.78 (0.28)
Statistical Analysis 1: Comparison: LY2196044 vs Placebo; Test type: Superiority or Other; p = 0.392, Mixed Models Analysis; Mean Difference (Final Values) = -0.32, 95% CI 2-sided [-1.05 to 0.41]

12. Secondary Outcome: Change From Baseline in Beck Anxiety Inventory (BAI) Total Score at Week 16 Endpoint
Description: BAI is a 21-item patient-completed questionnaire designed to assess the characteristics of anxiety. Participant was asked to rate how much he or she has been bothered by each symptom over the past week. Each item is rated on a 4-point scale (0=not present; 3=present in the extreme). Total scores range from 0 to 63. The higher the score, the more severe the anxiety symptoms. LS Mean value was controlled for treatment, pooled investigator, gender, family history, visit, baseline, gender*family history, treatment*visit, baseline*visit. An unstructured covariance structure was used.
Time Frame: Baseline, Week 16
Population: Participants with a baseline and post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2196044 | Placebo
Number analyzed (Participants) | 150 | 136
units on a scale | -1.98 (0.25) | -1.54 (0.26)
Statistical Analysis 1: Comparison: LY2196044 vs Placebo; Test type: Superiority or Other; p = 0.185, Mixed Models Analysis; Mean Difference (Final Values) = -0.44, 95% CI 2-sided [-1.10 to 0.21]

13. Secondary Outcome: Change From Baseline in Barratt Impulsivity Scale-11 (BIS-11) Total Score at Week 16 Endpoint
Description: The BIS-11 is a 30-item, self-administered impulsivity scale. Motor, cognitive, and non-planning domains are assessed and a total score is computed. This scale has previously been used in substance-abusing populations. Total scores range from 30-120. Higher scores indicate greater severity of symptoms. Least Squares (LS) Mean value was controlled for treatment, pooled investigator, gender, family history, baseline, gender*family history.
Time Frame: Baseline, Week 16
Population: Participants with a baseline and post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2196044 | Placebo
Number analyzed (Participants) | 120 | 99
units on a scale | -1.70 (0.65) | -2.95 (0.69)
Statistical Analysis 1: Comparison: LY2196044 vs Placebo; Test type: Superiority or Other; p = 0.142, ANCOVA; Mean Difference (Final Values) = 1.25, 95% CI 2-sided [-0.42 to 2.92]

14. Secondary Outcome: Change From Baseline in Thoughts About Abstinence Scale at Week 16 Endpoint
Description: Thoughts About Abstinence Scale was to measure participant's commitment to abstinence. It includes 3 items on a scale of 1-10: own desire to stop drinking (1=no desire to quit); own expectation of success in quitting (1=lowest expectation of success); how difficult to quit and remain abstinent (1=lowest amount of difficulty); and their goal related to alcohol use (scale of 1-7: 1=having no goal, up to total abstinence at 6 [7 was none of 6 above]). Least Squares (LS) Mean value was controlled for treatment, pooled investigator, gender, family history, baseline, gender*family history.
Time Frame: Baseline, Week 16
Population: Participants with a baseline and post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2196044 | Placebo
Number analyzed (Participants) | 123 | 100
units on a scale
  Desire to stop drinking at this time | -0.60 (0.20) | -0.11 (0.21)
  Expectation of success in quitting alcohol | -0.20 (0.25) | -0.00 (0.27)
  Difficulty to quit and remain abstinent | -1.11 (0.28) | -0.63 (0.30)
  Goal related to alcohol use | 0.00 (0.17) | 0.04 (0.18)
Statistical Analysis 1: Comparison: LY2196044 vs Placebo; Test type: Superiority or Other; p = 0.69, ANCOVA — P-value is for desire to stop drinking at this time; Mean Difference (Final Values) = -0.48, 95% CI 2-sided [-1.01 to 0.04]
Statistical Analysis 2: Comparison: LY2196044 vs Placebo; Test type: Superiority or Other; p = 0.545, ANCOVA — P-value is for expectation of success in quitting alcohol; Mean Difference (Final Values) = -0.20, 95% CI 2-sided [-0.85 to 0.45]
Statistical Analysis 3: Comparison: LY2196044 vs Placebo; Test type: Superiority or Other; p = 0.190, ANCOVA — P-value is for difficulty to quit and remain abstinent; Mean Difference (Final Values) = -0.48, 95% CI 2-sided [-1.20 to 0.24]
Statistical Analysis 4: Comparison: LY2196044 vs Placebo; Test type: Superiority or Other; p = 0.856, ANCOVA — P-value is for goal related to alcohol use; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.49 to 0.40]

15. Secondary Outcome: Change From Baseline in Quality of Life Enjoyment and Satisfaction Questionnaire Short Form (Q-LES-Q-SF) Total Score at Week 16 Endpoint
Description: Q-LES-Q-SF is a self-report instrument that assesses the degree of enjoyment and satisfaction in daily life activities. The domains include: social relationships, living or house situation, and physical health. Total scores range from 14-70. Higher scores indicate better quality of life. Least Squares (LS) Mean value was controlled for treatment, pooled investigator, gender, family history, visit, baseline, gender*family history, treatment*visit, baseline*visit. An unstructured covariance structure was used.
Time Frame: Baseline, Week 16
Population: Participants with a baseline and post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2196044 | Placebo
Number analyzed (Participants) | 150 | 133
units on a scale | 2.85 (0.56) | 2.08 (0.59)
Statistical Analysis 1: Comparison: LY2196044 vs Placebo; Test type: Superiority or Other; p = 0.297, Mixed Models Analysis; Mean Difference (Final Values) = 0.77, 95% CI 2-sided [-0.68 to 2.22]

16. Secondary Outcome: Change From Baseline in Endicott Work Productivity Scale (EWPS) Total Score at Week 16 Endpoint
Description: EWPS is a self-rated work productivity scale that assesses such topics as work hours, work missed, and behaviors and feelings related to the workplace. The EWPS will be completed only by subjects who work outside the home. There are 25 items and total scores range from 0-100. Higher scores indicate poorer productivity. Least Squares (LS) Mean value was controlled for treatment, pooled investigator, gender, family history, visit, baseline, gender*family history, treatment*visit, baseline*visit. An unstructured covariance structure was used.
Time Frame: Baseline, Week 16
Population: Participants with a baseline and post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2196044 | Placebo
Number analyzed (Participants) | 119 | 106
units on a scale | -5.67 (0.76) | -6.13 (0.79)
Statistical Analysis 1: Comparison: LY2196044 vs Placebo; Test type: Superiority or Other; p = 0.633, Mixed Models Analysis; Mean Difference (Final Values) = 0.46, 95% CI 2-sided [-1.44 to 2.36]

17. Secondary Outcome: Population Pharmacokinetic (PK) - Apparent Clearance
Description: Plasma concentrations were analyzed using population PK methodology with non-linear mixed effect modeling (NONMEM) software.
Time Frame: Over 16 weeks
Population: Participants who took study drug and contributed PK sample.
Measure: Mean (Standard Error); unit: Liter/hour (L/hr)
Groups:
- LY2196044: 250 milligram (mg) (titrate via 1 week at 50 mg and 1 week at 125 mg), once daily (QD), orally (PO), 16 weeks
Arm/Group | LY2196044
Number analyzed (Participants) | 169
Liter/hour (L/hr) | 36.5 (3.97)

18. Secondary Outcome: Population Pharmacokinetic (PK) - Apparent Volume of Distribution
Description: as for outcome 17
Time Frame: Over 16 weeks
Population: Participants who took study drug and contributed PK sample.
Measure: Mean (Standard Error); unit: Liter (L)
Arm/Group | LY2196044
Number analyzed (Participants) | 169
Liter (L) | 587 (8.38)

19. Secondary Outcome: Change From Baseline in Supine Blood Pressure (BP) at Week 16 Endpoint
Description: Least Squares (LS) Mean value was controlled for treatment, pooled investigator, visit, baseline, treatment*visit. An unstructured covariance structure was used.
Time Frame: Baseline, Week 16
Population: Participants who took at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: millimeters of mercury (mmHg)
Arm/Group | LY2196044 | Placebo
Number analyzed (Participants) | 186 | 179
millimeters of mercury (mmHg)
  Supine Systolic BP | -1.22 (0.68) | -0.45 (0.69)
  Supine Diastolic BP | -1.53 (0.43) | -1.08 (0.44)
Statistical Analysis 1: Comparison: LY2196044 vs Placebo; Test type: Superiority or Other; p = 0.409, Mixed Models Analysis — P-value is for supine systolic blood pressure; Mean Difference (Final Values) = -0.77, 95% CI 2-sided [-2.62 to 1.07]
Statistical Analysis 2: Comparison: LY2196044 vs Placebo; Test type: Superiority or Other; p = 0.452, Mixed Models Analysis — P-value is for supine diastolic blood pressure; Mean Difference (Final Values) = -0.45, 95% CI 2-sided [-1.63 to 0.73]

20. Secondary Outcome: Change From Baseline in Supine Pulse Rate at Week 16 Endpoint
Description: as for outcome 19
Time Frame: Baseline, Week 16
Population: Participants who took at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: beats per minute (bpm)
Arm/Group | LY2196044 | Placebo
Number analyzed (Participants) | 186 | 179
beats per minute (bpm) | -0.16 (0.51) | 0.37 (0.53)
Statistical Analysis 1: Comparison: LY2196044 vs Placebo; Test type: Superiority or Other; p = 0.456, Mixed Models Analysis; Mean Difference (Final Values) = -0.53, 95% CI 2-sided [-1.93 to 0.87]

21. Secondary Outcome: Change From Baseline in QTc Fridericia's Correction Interval (QTcF) Measured by Electrocardiograms at Week 16 Endpoint
Description: as for outcome 19
Time Frame: Baseline, Week 16
Population: Participants who took at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: milliseconds
Arm/Group | LY2196044 | Placebo
Number analyzed (Participants) | 148 | 135
milliseconds | -1.90 (0.86) | 0.18 (0.90)
Statistical Analysis 1: Comparison: LY2196044 vs Placebo; Test type: Superiority or Other; p = 0.081, Mixed Models Analysis; Mean Difference (Final Values) = -2.08, 95% CI 2-sided [-4.41 to 0.26]

22. Secondary Outcome: Percentage of Participants Discontinuation Due to Adverse Events (AEs)
Description: Percentage of participants discontinued study due to one or more AEs.
Time Frame: Baseline through Week 16
Population: Participants who took at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | LY2196044 | Placebo
Number analyzed (Participants) | 187 | 188
percentage of participants | 7.5 | 3.7
Statistical Analysis 1: Comparison: LY2196044 vs Placebo; Test type: Superiority or Other; p = 0.122, Fisher Exact

23. Secondary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (TEAE)
Description: Percentage of participants had one or more TEAEs during treatment period. TEAE is a worsening or new occurrence of adverse event during treatment compared to baseline.
Time Frame: Baseline through Week 16
Population: Participants who took at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | LY2196044 | Placebo
Number analyzed (Participants) | 187 | 188
percentage of participants | 76.5 | 61.7
Statistical Analysis 1: Comparison: LY2196044 vs Placebo; Test type: Superiority or Other; p = 0.002, Fisher Exact

24. Secondary Outcome: Change From Baseline in Orthostatic Blood Pressure (BP) at Week 16 Endpoint
Description: Orthostatic BP is the BP measured within 3 minutes of standing. Least Squares (LS) Mean value was controlled for treatment, pooled investigator, visit, baseline, treatment*visit. An unstructured covariance structure was used.
Time Frame: Baseline, Week 16
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | LY2196044 | Placebo
Number analyzed (Participants) | 186 | 179
mmHg
  Orthostatic Systolic BP | -1.23 (0.42) | -0.55 (0.43)
  Orthostatic Diastolic BP | -0.07 (0.27) | 0.25 (0.28)
Statistical Analysis 1: Comparison: LY2196044 vs Placebo; Test type: Superiority or Other; p = 0.235, Mixed Models Analysis — P-value is for orthostatic systolic blood pressure; Mean Difference (Final Values) = -0.69, 95% CI 2-sided [-1.82 to 0.45]
Statistical Analysis 2: Comparison: LY2196044 vs Placebo; Test type: Superiority or Other; p = 0.400, Mixed Models Analysis — P-value is for orthostatic diastolic blood pressure; Mean Difference (Final Values) = -0.31, 95% CI 2-sided [-1.05 to 0.42]

25. Secondary Outcome: Change From Baseline in Orthostatic Pulse Rate at Week 16 Endpoint
Description: Orthostatic pulse rate is the pulse rate measured within 3 minutes of standing. Least Squares (LS) Mean value was controlled for treatment, pooled investigator, visit, baseline, treatment*visit. An unstructured covariance structure was used.
Time Frame: Baseline, Week 16
Population: Participants who took at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: beats per minute
Arm/Group | LY2196044 | Placebo
Number analyzed (Participants) | 186 | 179
beats per minute | 0.65 (0.30) | -0.09 (0.31)
Statistical Analysis 1: Comparison: LY2196044 vs Placebo; Test type: Superiority or Other; p = 0.077, Mixed Models Analysis; Mean Difference (Final Values) = 0.74, 95% CI 2-sided [-0.08 to 1.57]

26. Secondary Outcome: Number of Participants With Clinical Institute Withdrawal Assessment for Alcohol Scale (CIWA-Ar)≥10 at Any Time From Baseline Through Week 16 Endpoint
Description: The revised CIWA-Ar scale measured the severity of alcohol withdrawal by rating 10 signs and symptoms: nausea; tremor; autonomic hyperactivity; anxiety; agitation; tactile, visual, and auditory disturbances; headache; and disorientation. Total scores range from 0-67. Higher scores indicate greater severity of withdrawal.
Time Frame: Baseline through Week 16
Population: Participants who took at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | LY2196044 | Placebo
Number analyzed (Participants) | 187 | 188
participants | 0 | 0

27. Secondary Outcome: Change From Baseline in Gastrointestinal Symptom Rating Scale (GSRS) Total Score at Week 16 Endpoint
Description: The GSRS is a clinician-administered scale used to assess upper and lower gastrointestinal physical symptoms. 15 items covering domains of abdominal pain, reflux syndrome, indigestion syndrome, diarrhea syndrome, and constipation syndrome were assessed with a 1-week recall period. Total scores range from 0-45. Higher scores indicate greater severity of symptoms. Least Squares (LS) Mean value was controlled for treatment, pooled investigator, gender, family history, visit, baseline, gender*family history, treatment*visit, baseline*visit. An unstructured covariance structure was used.
Time Frame: Baseline, Week 16
Population: Participants with a baseline and post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2196044 | Placebo
Number analyzed (Participants) | 185 | 179
units on a scale | 0.03 (0.13) | -0.54 (0.13)
Statistical Analysis 1: Comparison: LY2196044 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.57, 95% CI 2-sided [0.24 to 0.90]

ADVERSE EVENTS:
Groups:
- Placebo: once daily (QD), orally (PO), 16 weeks
Arm/Group | LY2196044 | Placebo
Serious Adverse Events (participants affected / at risk) | 4/187 | 5/188
Other Adverse Events (participants affected / at risk) | 143/187 | 116/188
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2196044 (N=187) | Placebo (N=188)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1)
Blood creatine phosphokinase mb increased (Investigations) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Alcoholism (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Alcohol detoxification (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2196044 (N=187) | Placebo (N=188)
Abdominal distension (Gastrointestinal disorders) | 12 (12) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 19 (22) | 6 (6)
Abdominal pain upper (Gastrointestinal disorders) | 11 (13) | 3 (4)
Constipation (Gastrointestinal disorders) | 12 (13) | 3 (5)
Diarrhoea (Gastrointestinal disorders) | 36 (39) | 16 (17)
Dyspepsia (Gastrointestinal disorders) | 6 (6) | 10 (11)
Flatulence (Gastrointestinal disorders) | 17 (17) | 9 (9)
Frequent bowel movements (Gastrointestinal disorders) | 8 (8) | 1 (1)
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 7 (8) | 3 (3)
Nausea (Gastrointestinal disorders) | 25 (28) | 12 (12)
Vomiting (Gastrointestinal disorders) | 11 (11) | 3 (3)
Fatigue (General disorders) | 17 (20) | 9 (9)
Upper respiratory tract infection (Infections and infestations) | 10 (11) | 7 (7)
Blood creatine phosphokinase increased (Investigations) | 4 (4) | 6 (9)
Decreased appetite (Metabolism and nutrition disorders) | 9 (10) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 7 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (9) | 7 (10)
Headache (Nervous system disorders) | 11 (17) | 17 (20)
Somnolence (Nervous system disorders) | 6 (6) | 2 (2)
Anxiety (Psychiatric disorders) | 6 (7) | 2 (2)
Libido decreased (Psychiatric disorders) | 6 (6) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 1 (1)
Hypertension (Vascular disorders) | 6 (6) | 3 (3)

LIMITATIONS AND CAVEATS:
Based on exposure data from an Alcohol Interaction study, H9T-MC-NABL (unregistered Phase 1 trial), the maximum dose in this study was reduced from 250 mg to 125 mg of LY2196044 after about 2/3 into the conduct of the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days